CLINICAL TRIAL: NCT03580993
Title: Ultrasonographic Evaluation of Lung and Heart in Predicting Successful Weaning in Mechanically Ventilated Neurosurgical Patients
Brief Title: Lung and Heart USG for Predicting Weaning in Neurosurgical Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health and Neuro Sciences, India (Other)
Responsible Party: Principal Investigator, Dhritiman Chakrabarti, Assistant Professor, National Institute of Mental Health and Neuro Sciences, India
Other Study IDs: IEC(BS & NS DIV)/2017-18
Record Dates: First submitted 2018-06-22; First posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Neurosurgery; Mechanical Ventilation; Extubation
Keywords: Critical Illness; Ultrasonography
MeSH Terms: conditions — Critical Illness | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SBT Completers: Those patients who successfully complete a spontaneous breathing trial of 2 hours.
  Interventions: Diagnostic Test: Lung Ultrasound
- SBT Non-completers: Those patients who fail to complete a spontaneous breathing trial of 2 hours.
  Interventions: Diagnostic Test: Lung Ultrasound

INTERVENTIONS:
Diagnostic Test: Lung Ultrasound — Lung ultrasound and Echocardiography used to derive parameters for prediction of successful SBT.
  Other Names: Echocardiography

SUMMARY:
Ultrasonography is a commonly used diagnostic and procedural adjunctive modality in intensive care. Weaning of neurosurgical patients off ventilatory support is a critical procedure, fraught with risks of hypoxia and hypercapnia. Weaning involves sequential reduction of ventilatory support and regular assessments for extubation followed by spontaneous breathing trials.

In this study, we evaluate parameters of ultrasonographic evaluation of lung aeration and cardiac function in neurosurgical patients undergoing weaning and their ability to predict successful weaning and extubation.

DETAILED DESCRIPTION:
Ultrasonography has become a ubiquitous feature of Intensive care nowadays, with its influence ranging from various diagnostics to various therapeutic interventions. It is readily available at the bedside and is non-invasive, making it an ideal tool in the hands of the intensivist. It has excellent safety profile, and hence can be performed repeatedly. These days it has become an indispensable tool in the intensive care units owing to its potential utility in the process of weaning a critically ill patient from mechanical ventilator support.

A neurosurgical patient is different from any other post-operative or critically ill patients. Their altered cerebral physiology, specific goals of therapy, varied response to usual management protocols, put them in a different league whole together. The primary aim of care for these patients is to detect and prevent any secondary neurological insult while supporting systemic and neurological homeostasis. Hypoxia and hypercarbia are factors which need to be absolutely avoided while caring for such patients. A good proportion of these patients will have respiratory instability, airway compromise and altered sensorium, which makes them prone to hypoxia and hypercarbia. To avoid these secondary insults to the neurological system, endotracheal intubation and mechanical ventilation is instituted in patients who are at high risk. Mechanical ventilation is continued until the patient is clinically stabilized and primary neurological damage has been taken care of. Subsequently the transition from control ventilation to spontaneous ventilation begins

The weaning process from mechanical ventilation involves sequential reduction of ventilatory parameters, assessment of readiness of the patient for extubation and when all these criterias are acceptable, then finally extubation. Daily, meticulous evaluation of clinical and neurological conditions and completion of spontaneous breathing trial (SBT) should be considered in order to recognize and facilitate the process of withdrawal of the mechanical ventilation. Extubation is considered as a success when the ventilator prosthesis is removed after the patient passed the SBT and there is no need for reinstitution of the MV in the next 48 hours. The entire process of weaning can be categorised as a six step process:

1. Taking care of the primary event
2. Deciding whether to start weaning
3. Assessing the readiness to wean
4. Spontaneous breathing trial (SBT)
5. Extubation
6. Assessment of probable reintubation6

Several parameters have been instituted for assessing the capability of weaning. These include: Rapid Shallow Breathing Index, which is the ratio of respiratory frequency to tidal volume (RSBI=f/VT), Pulmonary gas exchange (like: PaO2/FiO2, PaCO2), Vital Capacity (VC), Minute Ventilation and Static Compliance. Weaning may not always have a successful outcome. Difficult weaning may in fact be due to different or mixed etiologies, the diagnosis of which requires meticulous monitoring of various physiologic and objective parameters. Assessment of lung aeration by ultrasonography is rapidly gaining significance in weaning protocol. Apart from lung ultrasonography, the role of transthoracic echocardiography in successfully predicting weaning capability have been investigated in the recent times. Cardiac related weaning failure may be due to systolic LV dysfunction or isolated diastolic dysfunction. By this study we are trying to evaluate the scope of ultrasonography in detection of lung aeration and cardiac systolic and diastolic function in mechanically ventilated neurosurgical patients undergoing weaning; and whether they can be used as a good diagnostic tool to detect those who are likely to fail weaning in this specific subset of patient population.

ELIGIBILITY:
Inclusion Criteria:

1. All neurosurgical patients mechanically ventilated for more than 48 hrs and planned for weaning.
2. All patients whose underlying disease that required intubation was considered reversed or stabilised by the attending physician, rendering them eligible for spontaneous breathing trials.

Exclusion Criteria:

1. Uncooperative patient or the absence of a proper ultrasonographic window
2. Pregnancy
3. Patients having a GCS score of less than 8
4. Those having a pre weaning PaO2/ FiO2 ratio of less than 200
5. Severe ICU acquired neuromyopathy
6. Patients with lower cranial nerve involvement
7. Tracheostomised patients
8. Patients having high spinal cord lesions (above T8)
9. Presence of thoracostomy, pneumothorax or pneumomediastinum
10. Presence of rib fractures
11. Presence of pleural effusion
12. Patients having severe left ventricular dysfunction (LVEF < 35%)
13. Patients with planned prophylactic noninvasive ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neurosurgical patients being mechanically ventilated in ICU, being weaned off mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Change in Lung Ultrasound Score over the four study time points | Pre-SBT, Half hour during SBT, 2 hours during SBT, Pre-Extubation
  Each intercostal space of upper and lower parts of the anterior, lateral, and posterior regions of the left and right chest wall are carefully examined for four lung aeration patterns:
  1. Normal aeration
  2. Moderate loss of lung aeration
  3. Severe loss of lung aeration
  4. Lung consolidation
  For a given region of interest, points are allocated according to the worst ultrasound pattern observed: N = 0, B1 lines = 1, B2 lines = 2, C = 3. The LUS score ranging between 0 and 36 will be calculated as the sum of points.

SECONDARY OUTCOMES:
Change in Fractional Area Change over the four study time points | Pre-SBT, Half hour during SBT, 2 hours during SBT, Pre-Extubation
  Echocardiographic parameter measuring ventricular systolic function.
Change in Deceleration time of E over the four study time points | Pre-SBT, Half hour during SBT, 2 hours during SBT, Pre-Extubation
  Echocardiographic parameter measuring ventricular diastolic function.
Change in E:A Ratio over the four study time points | Pre-SBT, Half hour during SBT, 2 hours during SBT, Pre-Extubation
  Echocardiographic parameter measuring ventricular diastolic function.
Change in E:E' Ratio over the four study time points | Pre-SBT, Half hour during SBT, 2 hours during SBT, Pre-Extubation
  Echocardiographic parameter measuring ventricular diastolic function.
Change in Systolic Blood Pressure over the four study time points | Pre-SBT, Half hour during SBT, 2 hours during SBT, Pre-Extubation
  Systolic Blood Pressure
Change in Diastolic Blood Pressure over the four study time points | Pre-SBT, Half hour during SBT, 2 hours during SBT, Pre-Extubation
  Diastolic Blood Pressure
Change in Heart Rate over the four study time points | Pre-SBT, Half hour during SBT, 2 hours during SBT, Pre-Extubation
  Heart Rate

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Heath and Neurosciences, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No